CLINICAL TRIAL: NCT03252067
Title: Tear Concentrations and Pharmacokinetics of Azithromycin Following Topical Administration of a Single Dose of Azithromycin Eyedrops in Healthy Volunteers
Brief Title: Tear Concentrations and Pharmacokinetics of Azithromycin Eye Drops in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Grand Pharmaceutical (China) Co., Ltd. (Other)
Responsible Party: Principal Investigator, Xiuli Zhao, Prof., Beijing Tongren Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-PK-201402
Record Dates: First submitted 2017-08-04; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Pharmacokinetics
Keywords: Azithromycin eyedrops, pharmacokinetics, tears
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- azithromycin eyedrop (Experimental): Each of the subjects' eyes will receive single dose of azithromycin eyedrops and then attribute the time for tear sampling at seven time points up to 24 hours.
  Interventions: Drug: azithromycin eyedrop

INTERVENTIONS:
Drug: azithromycin eyedrop — Tear samples will be collected using the strips.

SUMMARY:
To evaluate azithromycin tear concentrations after one drop of azithromycin eyedrops (2.5ml/25mg) in healthy volunteers.

DETAILED DESCRIPTION:
In this randomized, open, single-center study, 42 healthy volunteers will receive one drop of azithromycin into each eye. Azithromycin tear concentrations will be measured by LC-MS/MS at seven time points for 24 hours. Tolerability is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old, male or female;
* BMI in the range of 19 to 24;
* eyes corrected visual acuity should be ≥ 1.0, intraocular pressure, slit lamp and fundus examination were normal, tear secretion function is normal;
* Good compliance and voluntarily signed consent.

Exclusion Criteria:

* Have eye disease or systemic disease;
* physical examination, laboratory tests, ECG and chest X-ray examination abnormalities and has clinical significance;
* HBsAg, anti-HCV, anti-HIV and TPPA positive;
* those who used eye drops two weeks before the test and who used any dosage form of azithromycin;
* known to azithromycin or macrolide-related varieties of allergies or serious adverse reactions;
* need to wear contact lenses during the test;
* history of internal surgery or laser surgery history;
* participated in other drug clinical trials in the past three months;
* pregnant women and lactating women, or in the growth period without taking effective contraceptive measures, menstrual period women;
* mental illness or alcohol, history of drug abuse or inability to collaborate;
* Any other circumstances that the investigators consider are unfit to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
the maximum concentration (Cmax) | The tear samples are taken at 7 time points after administration,including 10 minutes,half hour,2 hours,4 hours,8 hours,12 hours and 24hours.
  The tear samples are taken at 7 time points after administration up to 24 hours.The Cmax is calculated at the average concentration of each point.
area under the curve (AUC) | The tear samples are taken at 7 time points after administration,including 10 minutes,half hour,2 hours,4 hours,8 hours,12 hours and 24hours.
  The tear samples are taken at 7 time points after administration up to 24 hours.The AUC is calculated at the average concentration of each point.

SECONDARY OUTCOMES:
AEs | 24 hours
  Ocular and systemic adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No